CLINICAL TRIAL: NCT03015298
Title: Comparing the Diagnostic Role of 18F-FDG PET/MRI and of 18F-FDG PET/CT Among Patients With Gastric Cancer：A Randomized Controlled Trial
Brief Title: Comparing the Diagnostic Role of PET/MRI and of PET/CT Among Patients With Gastric Cancer
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Lin Chen, Director, Chinese PLA General Hospital
Other Study IDs: Experiment20160901
Record Dates: First submitted 2016-12-29; First posted 2017-01-10 (Estimated); Last update posted 2017-01-10 (Estimated); Status verified 2017-01

CONDITIONS: Gastric Cancer Stage
Keywords: gastric cancer; Simultaneous PET/MRI; PET/CT
MeSH Terms: conditions — Stomach Neoplasms | interventions — Positron Emission Tomography Computed Tomography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Gastric cancer: Each patient will perform a PET/MRI examination,and in the next day,a PET/CT.All the examinations are performed before the operation.
  Interventions: Device: PET/MRI; Device: PET/CT

INTERVENTIONS:
Device: PET/MRI — The recruited patients will receive a PET/MRI examination to evaluation the stage and resectability of the cancer.
  Other Names: Positron emission tomography-magnetic resonance imaging
Device: PET/CT — At the next day of PET/MRI examination,A PET/CT examination will be performed.
  Other Names: Positron emission tomography-computed tomography

SUMMARY:
The results of PET/MRI and PET/CT in each recruited gastric cancer patients will be compared.

DETAILED DESCRIPTION:
A prospective comparison of PET/MRI and PET/CT for gastric cancer will be performed,to evaluate the value of PET/MRI in predicting the preoperative staging and resectability of gastric cancer and investigate the role of PET/MRI in gastric cancer diagnosis.The evaluation parameters are the diagnostic accuracy of gastric cancer staging( including the overall accuracy, sensitivity, and specificity) and the receiver operating characteristic (ROC).

ELIGIBILITY:
Inclusion Criteria:

1. Histological diagnosis of gastric cancer
2. No previous treatment history for gastric cancer
3. Without complications of obstruction,bleeding and so on
4. Without severe diabetes,the levels of blood glucose <6.2 mmol/L .
5. No cardiac pacemarker,never stimulator or other metal substitute materials in vivo.

Exclusion Criteria:

1. With other neoplastic disease.
2. Suffering acute inflammatory disease
3. History of chemo-radiotherapy
4. Suffering prostate hyperplasia,glaucoma

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The cohort will recruit from patients diagnosed as gastric cancer and treated in the Department of general surgery.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-01; Primary Completion 2017-12 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
The results of the PET/MRI and PET/CT examination | 3 days
  Two experienced radiologists independently assess the TNM staging of gastric cancer using preoperative PET/MRI and PET/CT images

SECONDARY OUTCOMES:
Histopathological diagnosis | 5 days
  including definitely T stage in Tx, number of regional lymph node metastasis,result of histologic subtypes of carcinoma,result of other cytological examination.
Results of CT/Endoscopic ultrasound(EUS) image | 3 days
  Experienced radiologists assess definitely T stage in Tx, number of regional lymph node metastasis,with or without distant metastasis.
Numerical values of Standard uptake value(SUV) | 3 days
  Standard uptake value(SUV) is defined as the ratio of the image derived radioactivity concentration and the whole body concentration of the injected radioactivity.
Apparent Diffusion Coefficient(ADC) | 3 days
  Apparent Diffusion Coefficient(ADC) will be measured using a curved Placement of region of interest(ROI) to include the high signal and be read out on ADC maps by Diffusion-weighted magnetic resonance imaging (DWI or DW-MRI) analysis software.
The expression level of Receptor tyrosine-protein kinase erbB-2(HER2) | 5 days
  Acquire from pathology results
The expression level of Receptors for vascular endothelial growth factor(VEGFR) | 5 days
  Acquire from pathology results
Follow-up data | at lest 6 months
  results of conventional imaging examination and tumor biomarkers examination.

CONTACTS AND LOCATIONS:
Overall Officials: Jianxin Cui, Doctor, Study Director — the Chinese PLA General Hospital; Yi Liu, Principal Investigator — the Chinese PLA General Hospital

IPD SHARING:
Plan to Share IPD: No